CLINICAL TRIAL: NCT03048331
Title: The Effect of Functional Electrical Stimulation (FES) in Tetraplegia Reconstructive Surgery of the Upper Limbs - A Pilot Study
Brief Title: Functional Electrical Stimulation (FES) and Reconstructive Tetraplegia Hand and Arm Surgery
Acronym: FES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit further study participants
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-06
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury Cervical
Keywords: Functional Electrical Stimulation; Tetraplegia; Reconstructive Hand Surgery
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Electrical Stimulation (Experimental): Before surgery, the donor muscle is stimulated via surface electrodes in a loaded position or against resistance 3 times a week for 30 minutes.
  After surgery, the patients receive the same standard therapy as the control group. The electrical stimulation is performed once a day in combination with standard therapy for 30 minutes against gravity or resistance or in a loaded position.
  Interventions: Device: Functional Electrical Stimulation
- Standard therapy (No Intervention): Postoperatively, 20 min passive and active movements of the hand or arm are applied manually by a therapist. Additionally, the patients actively perform the same exercises once a day for 20 min. The movements are based on a standardised post-surgical treatment protocol.

INTERVENTIONS:
Device: Functional Electrical Stimulation — Functional electrical stimulation is applied with stimulators according to the lesion. In case of a upper motor neuron lesion the stimulation operates via nerve. For the stimulation surface electrodes are placed on the skin over the muscle belly. The stimulation of the innervated muscles will be conducted using the following conditions:
  300-400 usec, 20-50 Hz, amplitude depends on the quality of muscle contraction (20-80 mA). the duty cycle of the stimulation is 3 sec. ramp up, 5 ec. plateau, 2 sec. ramp down, 10 sec. pause.
  Arms: Functional Electrical Stimulation

SUMMARY:
FES is a common and established method in the rehabilitation of persons with spinal cord injury (SCI). Some known effects of FES were investigated in several studies e.g. avoiding disuse and denervation atrophy, improving muscle force, power output and endurance changing muscle fibre type, increasing cross sectional area of muscle, increasing muscle mass, activation of nerve sprouting, reducing spasticity and motor learning.

Most of the studies investigated the impact of FES in the lower limbs. For the upper extremities fewer studies exist. However, it is supposed that the effects of FES are similar.

In the rehabilitation of persons with tetraplegia, FES, especially the stimulation of the upper extremities triggered by electromyography (EMG) is an established method to generally improve hand and arm function. However, none of those studies has investigated the effect of FES in combination with reconstructive tetraplegia hand surgery. Improved muscle strength is supposed to improve the functional outcome in participation. Additionally, FES could increase the motor learning process. Supported by the clinical observation we hypothesize that FES has a positive influence on the outcome of surgical reconstruction of tendon and/or nerve transfers.

DETAILED DESCRIPTION:
In the rehabilitation of patients with a tetraplegia, FES is a common used method to improve the function of the arms and hands. The effects of FES also gain in importance considering the procedure of reconstructive arm and/or hand surgery in tetraplegic patients. The functioning of arm and hand muscles can be improved by surgically inverting intact muscles. Therefore, strengthening of the donor and recipient muscles with FES seems to be reasonable. So far it is not established if systematic training with FES before and after reconstructive hand and arm surgery could additionally improve the outcome in terms of strength, motor learning and function. However, clinical observations show a possible positive effect of FES.

The aim of the present randomized controlled study is to evaluate the use of FES before and after a reconstructive arm and/or hand surgery in order to increase the strength of the donor and recipient muscles, and thus, improving the result regarding strength and functionality.

A total of 30 tetraplegic patients who are planned to have a reconstructive arm and/or hand surgery at the Swiss Paraplegic Centre will be included into the study. The participating subjects will be randomized into two groups: a control and an intervention group.

The control group (15 patients) will receive defined standardized physio- and occupational therapy after the surgery. The intervention group (15 patients) will receive a combination of standardized physio- and occupational therapy and FES, before and after surgery. The standardized therapy will be supplemented with FES for 3 months, 3 x 30min per week.

To verify the effects of FES on muscular strength and functionality of the arms and hands, several assessments will be conducted at 4 different time points (T1: 12 weeks before surgery // T2: just before surgery // T3: 4 weeks post-surgery // T4: 16 weeks post-surgery). The course of the voluntary muscular strength and the strength generated by FES of both, the donor and the recipient muscle will be measured. In addition, the change in muscle volume in forearm and upper arm will be assessed by ultrasound. Furthermore, a standardized test to check several grasping action will be performed and there will also be a manual testing of the muscles in arms and hands.

Statistical analysis of these assessments enable an estimation of the benefit and effect of FES as an additional therapy in the context of reconstructive arm and/or hand surgery for tetraplegic patients.

ELIGIBILITY:
Inclusion Criteria:

* traumatic or non-traumatic (> 6 month) spinal cord injury
* Age ≥ 18 years
* Level of lesion C4 - Th1
* American Spinal Cord Injury Association Impairment Scale (AIS) A/B/C/D
* Planned reconstructive hand or arm surgery at the Swiss Paraplegic Centre Nottwil
* Signed informed consent

Exclusion Criteria:

* Patients during primary rehabilitation
* Patients' inability to follow the study, e.g. mental-health problems, language problems, dementia etc.
* Pregnancy (anamnestic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
Change in evoked force | 12 weeks before surgery, 1 day before surgery, 4 weeks post-surgery and 16 weeks post-surgery
  Change in voluntary and electro-stimulated evoked force (torque Nm) for the recipient muscle
Change in power output | 12 weeks before surgery, 1 day before surgery, 4 weeks post-surgery and 16 weeks post-surgery
  Change in voluntary and electro-stimulated power output (W) for the recipient muscle

SECONDARY OUTCOMES:
Change in Canadian Occupational Performance Measurement (COPM) | 2 weeks before surgery, 1 day before surgery and 16 weeks post-surgery
  Changes of functional outcomes (i.e. performance and satisfaction) of the treated upper limb before and after surgery
Change in muscle volume | 2 weeks before surgery, 1 day before surgery and 16 weeks post-surgery
  Difference in muscle volume of the treated limb before and after surgery measured by ultrasound
Change in the treatment effectiveness | 2 weeks before surgery, 1 day before surgery and 16 weeks post-surgery
  Questionnaire of the participant's perception of the treatment effectiveness to evaluate the benefit of FES according to effort of the treatment
Change in muscle activity | 4 weeks post-surgery and 16 weeks post-surgery
  Change in the muscle activity of a transferred muscle in a new function surface assessed by EMG

CONTACTS AND LOCATIONS:
Overall Officials: Jan Fridén, Prof. Dr. med., Principal Investigator — Swiss Paraplegic Centre Nottwil, Switzerland
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No